CLINICAL TRIAL: NCT00505700
Title: Phase I Dose Escalating Trial of VELCADE (PS-341) in Combination With Idarubicin and Cytosine Arabinoside in Patients With Acute Myelogenous Leukemia
Brief Title: VELCADE in Combination With Idarubicin and Cytosine Arabinoside in Patients With Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Philip Amrein, MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-103
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Leukemia
Keywords: acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Bortezomib; Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: velcade
Drug: Idarubicin
Drug: Cytarabine

SUMMARY:
The primary objective of this study is to establish the maximally tolerated dose of VELCADE that can be administered with idarubicin and cytarabine in patients with AML. The secondary objectives of this study are assessment of efficacy, safety, and pharmacokinetics of Velcade when combined with Cytarabine and idarubicin. Various molecular markers associated with response to Velcade, cytarabine, and idarubicin will be explored by utilizing microarray analyses. The study endpoints are maximum tolerated dose and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older.
* Unequivocal histologic diagnosis of AML (>20% blasts in the blood and/or bone marrow based on the WHO and/or FAB classifications as described in Appendix 9.3), excluding M3 (acute promyelocytic leukemia).
* For patients less than 60, disease must have previously achieved CR and then relapsed (>20% blasts in the blood and/or bone marrow based on the WHO and/or FAB classifications as described in Appendix 9.3), excluding M3 (acute promyelocytic leukemia).). These patients must have a period of remission of >3 months (beginning with the time when the ANC >1,500/ul, platelets >100,000/ul and < 5% marrow blasts are present).
* Patients 60 years of age or older may have relapsed disease or may have previously untreated AML (>20% blasts in the blood and/or bone marrow based on the WHO and/or FAB classifications as described in Appendix 9.3), excluding M3 (acute promyelocytic leukemia).
* Patients may have prior myelodysplasia. Patients may have prior treatment for myelodysplasia.
* Patients may have had prior chemotherapy for another malignancy or an antecedent hematologic disorder such as myelodysplasia.
* Patients must have an ECOG performance status 0-3.
* Patients must have all of the following pretreatment laboratory values within 21 days of enrollment: total bilirubin <= 1.5 X the upper limit of normal (ULN), ALT and AST <= 2.5 X the ULN, creatinine <= 2.0 mg/dl.
* Male patients need to use an appropriate method of barrier contraception during the study.
* Female patients must be post-menopausal, surgically sterilized, or willing to use acceptable methods of birth control (i.e. a hormonal contraceptive, an intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Patients must give voluntary written informed consent before performance of any study-related procedure not part of normal medical care.

Exclusion Criteria:

* If less than 60 years old, patient has received chemotherapy within the last three months (90 days).
* Patients with untreated AML < 60 years old.
* Other active malignancy (with the exception of basal and squamous cell skin cancer) at the time of study entry.
* Patient has hypersensitivity to boron or mannitol
* Severe pulmonary or cardiac disease.
* History of congestive heart failure or ejection fraction < 40%.
* Patient had a myocardial infarction within 6 months of enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Patients with M3 AML (acute promyelocytic leukemia) by FAB or WHO as described in 9.3.
* Patients with HIV infection.
* Patients with known active hepatitis B or C.
* Patients with known central nervous system leukemia. A lumbar puncture is not required unless CNS involvement is clinically suspected.
* Patients who are pregnant or breast feeding.
* Patients with major surgery within the 4 weeks prior to trial enrollment.
* Patients with ³ Grade 2 peripheral neuropathy within 21 days before enrollment.
* Patients with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia. If the condition becomes controlled, the patient may become eligible.
* Patients with any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2003-07; Primary Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip C Amrein, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel/ Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts